CLINICAL TRIAL: NCT07097610
Title: The Effect of Mosaic Puzzle Game on Nomophobia in Adolescents: A Randomised Controlled Study
Brief Title: The Effect of Mosaic Puzzle Game on Nomophobia in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabia Nur TEKİ KESKİN (Other)
Collaborators: Pamukkale University scientific research project department (Unknown)
Responsible Party: Sponsor-Investigator, Rabia Nur TEKİ KESKİN, Nurse (PhD Candidate), Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PamukkaleU-SBE-RNTK-01
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Nomophobia; Puzzle Activity; Child; Dependence; Smart Phone Addiction
Keywords: nomophobia; child; dependence; smart phone addiction; puzzle activity

STUDY DESIGN:
Intervention Model Description: The study includes one intervention group and one control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: "Mosaic Puzzle Intervention Group" (Experimental): Arm Description: In the study, the child's level of nomophobia will first be determined using a Personal Information Form and a nomophobia measurement tool. Subsequently, the mosaic puzzle intervention will be administered to the children in the experimental group twice a week for one hour over a period of five weeks, at times deemed appropriate by the school, and will be monitored by the researcher.
  Mosaic Puzzle Initiative A mosaic puzzle is the process of creating a picture or image by putting together small crystal stones. It involves sticking the appropriate crystal stones onto a canvas painting using wax and a wax pencil, matching them with the symbols (letters, numbers, shapes, etc.) shown on the painting. (e.g., sticking blue crystal stones gathered under the * symbol onto the square marked with * on the canvas). The student presses the wax pencil onto the wax to pick up a small amount of wax. Then, they press the wax-coated pencil onto the crystal stone and stick it onto the
  Interventions: Other: Mosaic Puzzle Intervention
- No Intervention: Control Group (No Intervention): Arm Description: In the study, the child's level of nomophobia will first be determined using the Personal Information Form and the Nomophobia measurement tool in the control group. No intervention will be performed on the children in this group, and a test will be administered at the end of the intervention.

INTERVENTIONS:
Other: Mosaic Puzzle Intervention — This study aims to investigate the effect of mosaic puzzle application on nomophobia in adolescents. The data for the study will be collected over a 5-week period. The experimental group children will be asked to play mosaic puzzle games for 1 hour, 2 days a week for 5 weeks at a time deemed appropriate by the school under the supervision of the researcher. The control group children will not be given any application; they will only be observed, and a final test will be administered at the end of the 5 weeks. The study is planned as a single-center study, and a total of 30 children aged 12-14 with a nomophobia scale score of 60 or higher who meet the inclusion criteria will be included in the study.
  Arms: Experimental: "Mosaic Puzzle Intervention Group"

SUMMARY:
This study aims to investigate the effect of mosaic puzzle application on nomophobia in middle school children aged 12-14.

The data for the study will be collected over a 5-week period. The experimental group children will be asked to play mosaic puzzle games for 1 hour, 2 days a week for 5 weeks, at a time deemed appropriate by the school and under the supervision of the researcher. The control group children will not be given any intervention; they will only be observed, and a final test will be administered at the end of the 5 weeks. The study is planned as a single-center study, and a total of 30 children aged 12-14 with a nomophobia scale score of 60 or higher who meet the inclusion criteria will be included in the study.

Hypothesis 1: The intervention group's level of nomophobia is lower than that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Score at least 60 points on the nomophobia scale
* Be between the ages of 12 and 14
* Written consent from parents and verbal consent from the child

Exclusion Criteria:

* Be under 12 years of age and over 14 years of age
* Have scored less than 60 points on the nomophobia scale

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Nomophobia Scale (NO) for the 9-18 Age Group | From enrollment to the end of treatment at 10 weeks.
  The Nomophobia Scale developed by Yıldırım and Correia (2015) is a Likert-type measure that assesses the level of fear experienced by children when they do not have access to their cell phones. The validity and reliability of the scale were studied by Özdemir and Bektaş (2020). The scale consists of 20 items. It is a 7-point Likert-type scale (1: Strongly disagree; 7: Strongly agree). The scale has four subscales: inability to access information, giving up comfort, inability to communicate, and loss of online connection. A score of 20 on the scale indicates no nomophobia, 21 ≤ NÖ Score < 60 indicates mild nomophobia, 60 ≤ NÖ Score < 100 indicates moderate nomophobia, and 100 ≤ NÖ Score ≤ 140 indicates severe nomophobia. The scale ranges from a minimum of 20 to a maximum of 140 points. As the score increases, the level of nomophobia increases. Individuals who score 61 or higher on the raw score can be classified as having 'severe or moderate' nomophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No